CLINICAL TRIAL: NCT04084301
Title: Impact of Cardiopulmonary Bypass Flow on Renal Oxygenation, Blood Flow and Tubular Injury
Acronym: ICAROX2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lukas Lannemyr, Specialist of Anesthesia and Intensive care, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICAROX2
Record Dates: First submitted 2019-02-04; First posted 2019-09-10 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Extracorporeal Circulation; Complications; Renal Failure; Circulation Disorder; Renal Plasma Flow, Effective; Cardiopulmonary Bypass; Hemolysis; Inflammatory Response
Keywords: renal oxygenation; renal blood flow; cardiopulmonary bypass; tubular cell injury; N-acetyl-beta-D-glucosaminidase; nephrocheck; inflammation; hemolysis
MeSH Terms: conditions — Renal Insufficiency; Hemolysis; Gangliosidoses, GM2; Inflammation

STUDY DESIGN:
Intervention Model Description: To compare normal (2.4 L/min/m2) and high (2.9 L/min/m2) cardiopulmonary bypass flow during cardiac surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal CPB flow (No Intervention): In this group, the target flow during cardiopulmonary bypass (CPB) will be 2.4 L/min/m2 throughout the CPB period.
- High CPB flow (Experimental): In this group, the target flow during cardiopulmonary bypass (CPB) will be 2.9 L/min/m2 throughout the CPB period.
  Interventions: Procedure: High CPB flow

INTERVENTIONS:
Procedure: High CPB flow — Target CPB flow 2.9 L/min/m2 throughout the CPB period
  Arms: High CPB flow

SUMMARY:
During open cardiac surgery, cardiopulmonary bypass (CPB) is used to temporarily replace the function of the heart and lungs. Renal ischemia resulting in acute kidney injury is common after cardiac surgery. The renal oxygenation is impaired during CPB, but the oxygenation may be improved by increasing the CPB blood flow. In this randomized study, two CPB flow rates will be compared regarding renal outcome (biomarkers and renal oxygenation/renal blood flow), as well as markers of inflammation and hemolysis. Additionally, urine oxygen tension will be measured during CPB and the early intensive care phase and compared to renal oxygenation. Regional oxygen saturation assessed with near infrared spectroscopy from the brain and kidneys will be monitored during and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed informed consent
* Male and female subjects ≥18 years
* Left ventricular ejection fraction ≥30 %
* Estimated GFR ≥30 ml/min using the CKD-EPI equation (Levey 2009)
* Scheduled open cardiac surgery with CPB
* Planned normothermia during CPB
* Expected CPB time > 60 minutes

Exclusion Criteria:

* Emergency surgery
* Cardiac transplantation
* Advanced grown-up congenital heart disease corrections
* Previous cerebral infarction, verified with computed tomography or magnetic resonance imaging
* Body mass index > 32 kg/m2
* Use of hypothermia < 32 °C during CPB
* Inability of the patient to give based opinion
* In the investigator´s opinion, the patient has a condition that could be adversely affected by study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Biomarker u-NAG | 24 hours
  Tubulus injury biomarker N-acetyl-ß-d-glucoseaminidase (NAG) will be analyzed in urine with a spectrophotometric method and corrected for urine creatinine.
Biomarkers Nephrocheck | 24 hours
  Renal biomarker assay Nephrocheck (IGFBP-7 x TIMP-2) will be analyzed in urine
Renal oxygen delivery and blood flow | 6 hours
  Renal oxygen delivery during and after cardiopulmonary bypass (CPB)

SECONDARY OUTCOMES:
Serum creatinine and acute kidney injury (AKI) | 48 hours
  Changes in serum creatinine
Inflammation IL-1 | 24 hours
  Differences in inflammatory marker IL-1
Inflammation IL-6 | 24 hours
  Differences in inflammatory marker IL-6
Inflammation IL-8 | 24 hours
  Differences in inflammatory marker IL-8
Inflammation IL-10 | 24 hours
  Differences in inflammatory markers IL-1, IL-6, IL-8, IL-10 and TNFa
Inflammation TNFa | 24 hours
  Differences in inflammatory marker TNFa
Complement activation | 24 hours
  Differences in complement activation
Hemolysis | 24 hours
  Differences in markers of hemolysis (free plasma Hb, LD, haptoglobin)
Erythropoetin | 24 hours
  Differences in serum-erythropoietin
Neuroinflammation Tau | 4 days
  Changes in Tau
Neuroinflammation NF | 4 days
  Changes Neurofilament
Kidney function | 24 hours
  Measured glomerular filtration rate (iohexol clearance) on postoperative day 1
Renal function | 24 hours
  Measured glomerular filtration rate by iohexole clearance on the first postoperative day

OTHER OUTCOMES:
Urinary pO2 | 24 hours
  Changes in urinary pO2 measured with laser doppler technique. Correlation with global renal oxygenation will be explored.

CONTACTS AND LOCATIONS:
Locations (1):
- Lukas Lannemyr, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lannemyr L, Bragadottir G, Krumbholz V, Redfors B, Sellgren J, Ricksten SE. Effects of Cardiopulmonary Bypass on Renal Perfusion, Filtration, and Oxygenation in Patients Undergoing Cardiac Surgery. Anesthesiology. 2017 Feb;126(2):205-213. doi: 10.1097/ALN.0000000000001461. PMID 27906706
- [Result] Lannemyr L, Bragadottir G, Hjarpe A, Redfors B, Ricksten SE. Impact of Cardiopulmonary Bypass Flow on Renal Oxygenation in Patients Undergoing Cardiac Operations. Ann Thorac Surg. 2019 Feb;107(2):505-511. doi: 10.1016/j.athoracsur.2018.08.085. Epub 2018 Oct 23. PMID 30365961
- [Result] Lannemyr L, Lundin E, Reinsfelt B, Bragadottir G, Redfors B, Oras J, Ricksten SE. Renal tubular injury during cardiopulmonary bypass as assessed by urinary release of N-acetyl-ss-D-glucosaminidase. Acta Anaesthesiol Scand. 2017 Oct;61(9):1075-1083. doi: 10.1111/aas.12946. Epub 2017 Jul 26. PMID 28748536